CLINICAL TRIAL: NCT01583374
Title: A PHASE 3, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY TO EVALUATE THE EFFICACY AND SAFETY OF APREMILAST (CC-10004) IN THE TREATMENT OF ACTIVE ANKYLOSING SPONDYLITIS
Brief Title: Study of Apremilast to Treat Subjects With Active Ankylosing Spondylitis
Acronym: POSTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CC-10004-AS-001; 2011-001555-37 (EudraCT Number)
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Ankylosing Spondyloarthritis
Keywords: spondylitis; spondyloarthritis; Spondyloarthropathy; Oral preparation
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylitis; Spondylarthritis; Spondylarthropathies | interventions — apremilast; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apremilast 20 mg (Experimental): Apremilast 20 mg was taken orally twice a day (BID)
  Interventions: Drug: Apremilast tablet 20 mg
- Apremilast 30 mg (Experimental): Apremilast 30 mg was taken orally twice a day
  Interventions: Drug: Apremilast tablet 30 mg BID
- Placebo (Placebo Comparator): Identically matched placebo tablets were taken orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast tablet 20 mg — Apremilast 20 mg was taken orally twice a day (BID)
  Other Names: Otezla; CC-10004
  Arms: Apremilast 20 mg
Drug: Apremilast tablet 30 mg BID — Apremilast 30 mg was taken orally twice a day
  Other Names: Otezla; CC-10004
  Arms: Apremilast 30 mg
Drug: Placebo — Identically matched placebo tablets were taken orally twice a day during the placebo controlled phase.
  Arms: Placebo

SUMMARY:
Apremilast is a new, orally available, small molecule drug that specifically inhibits phosphodiesterase 4 (PDE4), an enzyme that modulates inflammatory cytokines. This clinical study tests whether apremilast can improve the signs and symptoms of ankylosing spondylitis.

DETAILED DESCRIPTION:
Patients were randomized in a 1:1:1 ratio to placebo, apremilast 20 mg BID and apremilast 30 mg BID. The duration of the study was approximately 5 years. The double blind period (when patients nor the physician knew whether placebo or apremilast was taken) was 24 weeks. At Week 16, participants who did not have either a ≥ 20% improvement or a ≥ 1 unit improvement from baseline in at least two of the four SpondyloArthritis international Society (ASAS) domains were entered in "early escape" from their current treatment in a double-blinded manner. However, such participants were permitted to continue in the study. At Week 24, participants may have entered a long-term extension phase for up to an additional 4.5 years (236 weeks). At "second escape" (at Week 24), apremilast 20 mg BID treated participants transitioned to receive double-blinded apremilast 30 mg BID and remained on double-blinded apremilast 30 mg BID because they continued to improve with a longer duration of treatment. After Week 24 and during the early portion of the long-term extension through Week 52, all participants continued on either double-blinded apremilast 20 mg BID or 30 mg BID treatment. After all participants had completed Week 52 or had terminated early from the study and the 52-week data base was locked, apremilast 20 mg BID or 30 mg BID treatment was provided.

ELIGIBILITY:
Inclusion Criteria:

* Must have a documented diagnosis of ankylosing spondylitis as defined by low back pain and stiffness, which improves with exercise, but is not relieved by rest for more than 3 months prior to screening. At the completion of screening procedures, a documented diagnosis of definite active AS, as defined by the modified New York criteria (1984) whereby both criteria, at least 1 radiographic criterion and at least 1 clinical criterion, must be met
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is ≥ 4
* Total back pain is ≥ 4
* On stable dose of AS medication (or lack of medication) prior to randomization and through week 24

Exclusion Criteria:

- Prior treatment with a Tumor Necrosis Factor (TNF) blocker and any biologic treatment for AS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2014-02-24 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (103):
- United States (20):
  - Sun Valley Arthritis Center, Peoria, Arizona
  - University of California, San Diego, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - UCSF Arthritis Center, San Francisco, California
  - Advent Clinical Research Centers, Inc, Pinellas Park, Florida
  - Burnette & Silverfield, MDS PLC, Tampa, Florida
  - Alastair Kennedy, MD Research, Vero Beach, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Saint Paul Rheumatology, PA, Eagan, Minnesota
  - MetroHealth Medical Systems, Cleveland, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Arthritis Clinic, Jackson, Tennessee
  - Ramesh C Gupta MD, Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Australia (5):
  - Southern Clinical Research, Hobart, Tasmania
  - Emeritus Research, Camberwell, Victoria
  - Coastal Joint Care, Maroochydore
  - Royal Perth Hospital, Perth
  - The Queen Elizabeth Hospital, Woodville South
- Krankenhaus Wien-Hietzing, Vienna, Austria
- Bulgaria (5):
  - Diagnostic and Consulting Center Sv. Pantaleymon, Pleven
  - National Multiprofile Transport Hospital Tzar Boris III, Sofia
  - 17 Diagnostic and Consulting Centre, Sofia
  - Military Medical Academy - MHAT, Sofia
  - Diagnostic Consulting Center N4, Varna
- Canada (9):
  - Clinic: University of Calgary Heritage Medical Research Clinic (HMRC),Teaching Research and Wellness (TRW), Calgary, Alberta
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Cividino Medicine Professional Corporation, Hamilton, Ontario
  - Dr. William G. Bensen Medicine Professional Corporation, Hamilton, Ontario
  - Credit Valley Professional Building, Mississauga, Ontario
  - The Arthritis Program Research Group Inc., Newmarket, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Saint-Louis, Quebec
- Czechia (8):
  - Revmatologie s.r.o., Brno
  - ARTMEDI UPD s.r.o., Hostivice
  - ARTHROMED s.r.o., Pardubice
  - Revmatologicka Ambulance, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou - Klinicko-farmakologicka jednotka, Prague
  - Medifin a.s, Šustova, Prague
  - Revmatologicka Ambulance, Sokolov
  - PV-Medical s.r.o., Zlín
- Estonia (4):
  - Innomedica Medical and Research Centre, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - Clinical Research Centre Ltd, Tartu
  - Tartu University Hospital, Tartu
- France (5):
  - Hopital Ambroise-Pare, Boulogne
  - Hopital Henri Mondor, Créteil
  - IPROS - CHR ORLEANS - Hôpital de la Source, Orléans
  - Hopital Cochin, Paris
  - Groupe Hospitalier Pitié- Salpétrière, Paris
- Germany (6):
  - Charite - Universitätsmedizin Berlin, Berlin
  - Universitatsklinikum Erlangen, Erlangen
  - Centrum fur innovative Diagnostik und Therapie Rheumatologie Immunologie GmbH, Frankfurt
  - Schön Klink Hamburg-Eilbek, Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Rheumazentrum Ruhrgebiet, Herne
- Hungary (5):
  - Qualiclinic kft, Budapest
  - Synexus Magyarország Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Veszprem Megyei Csolnoky Ferenc Korhaz-Rendelointezet, Veszprém
- Netherlands (2):
  - Leiden Universitair Medisch Centrum, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
- Poland (8):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - NZOZ Osteo-Medic sc A. Racewicz J. Supronik, Bialystok
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Synexus SCM Sp. z o.o., Gdynia
  - Zespol Poradni Specjalistycznych, Lublin
  - Prywatna Praktyka Lekarska Pawel Hrycaj, Poznan
  - NZOZ NASZ LEKARZ Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna, Torun
  - Synexus SCM Sp. z o.o., Wroclaw
- Romania (5):
  - Cristei R. Rodica - Private Medical Practice, Brăila
  - Sf. Maria Clinical Hospital, Bucharest
  - Emergency County Clinical Hospital, Cluj-Napoca
  - Sf Apostol Andrei Emergency Clinical County Hospital, Galati
  - RK Medcenter SRL, Iași
- Russia (7):
  - Research Medical Complex Vashe Zdorovie, Kazan'
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Federal State Budget Institution "Rheumatology Research Institute RAMS", Moscow
  - Nizhniy Novgorod State Medical Academy of Roszdrav, Nizhny Novgorod
  - Departmental Hospital at Smolensk Station RZhD JSC, Smolensk
  - Regional Clinical Hospital, Vladimir
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg
- Slovakia (2):
  - Narodny ustav reumatickych chorob, Piešťany
  - MUDr. Zuzana Cizmarikova, s.r.o., Reumatologick ambulancia, Poprad
- Spain (6):
  - Hospital Universitario a Coruna, A Coruña
  - Hospital de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Corporacio Sanitaria Parc Tauli de Sabadell, Sabadell
  - Complejo Hospitalario Universitario de Santiago de Compostela Travesía de la Choupana s/n, Santiago de Compostela
- Skånes Universitetssjukhus- Malmö, Malmo, Sweden
- United Kingdom (4):
  - Barnsley Hospital, Barnsley
  - Royal National Hospital for Rheumatic Diseases, Bath
  - Chapel Allerton Hospital, Leeds
  - Nuffield Orthopaedic Centre, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Gladman DD, Kavanaugh A, Gomez-Reino JJ, Wollenhaupt J, Cutolo M, Schett G, Lespessailles E, Guerette B, Delev N, Teng L, Edwards CJ, Birbara CA, Mease PJ. Therapeutic benefit of apremilast on enthesitis and dactylitis in patients with psoriatic arthritis: a pooled analysis of the PALACE 1-3 studies. RMD Open. 2018 Jun 27;4(1):e000669. doi: 10.1136/rmdopen-2018-000669. eCollection 2018. PMID 30018799
- [Background] Kavanaugh A, Gladman DD, Edwards CJ, Schett G, Guerette B, Delev N, Teng L, Paris M, Mease PJ. Long-term experience with apremilast in patients with psoriatic arthritis: 5-year results from a PALACE 1-3 pooled analysis. Arthritis Res Ther. 2019 May 10;21(1):118. doi: 10.1186/s13075-019-1901-3. PMID 31077258
- [Derived] Taylor PC, van der Heijde D, Landewe R, McCue S, Cheng S, Boonen A. A Phase III Randomized Study of Apremilast, an Oral Phosphodiesterase 4 Inhibitor, for Active Ankylosing Spondylitis. J Rheumatol. 2021 Aug;48(8):1259-1267. doi: 10.3899/jrheum.201088. Epub 2021 Feb 15. PMID 33589554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants at 88 study sites and in 18 countries (Australia, Austria, Bulgaria, Czech Republic, Estonia, France, Germany, Hungary, the Netherlands, Poland, Romania, Russia, Slovakia, Spain, the United Kingdom, Canada, Sweden, and the United States [US]).
Pre-assignment Details: Randomized participants were stratified by the following 2 parameters:
  1. C-Reactive Protein (CRP) concentration (normal: ≤ 1.5 mg/dL or elevated: > 1.5 mg/dL) at screening;
  2. The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score < 6.0 or BASDAI score ≥ 6.0 at baseline.
Groups:
- Placebo: Participants initially randomized to receive placebo tablets BID in the 24-week placebo-controlled phase.
- Apremilast 20 mg: Participants initially randomized to 20 mg apremilast tablets BID in the 24-week placebo-controlled phase continued to receive 20 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
- Apremilast 30 mg: Participants initially randomized to 30 mg apremilast tablets BID in the 24-week placebo-controlled phase, continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
- Placebo / Apremilast 30 mg Early Escape (EE): Participants initially randomized to receive placebo tablets BID who did not have at least 20% improvement or ≥ 1 unit improvement from baseline in 2 out of 4 of the Assessment of SpondyloArthritis International Society (ASAS) domains at Week 16 were transitioned to 30 mg apremilast tablets BID and continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
- Placebo/Apremilast 30 mg Crossover (XO): Participants initially randomized to placebo tablets BID in the 24-week placebo controlled phase were transitioned to 30 mg apremilast tablets BID at Week 24 and continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
- Apremilast 30 mg /Apremilast 30 mg EE: Participants initially randomized to 30 mg apremilast tablets BID in the 24-week placebo-controlled phase who did not have at least 20% improvement or a ≥ 1-unit improvement from baseline in 2 of the 4 ASAS domains at Week 16 continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
- Apremilast 20 mg /Apremilast 30 mg EE: Participants initially randomized to 20 mg apremilast tablets BID who did not have at least 20% improvement or ≥ 1 unit improvement from baseline in 2 out of 4 of the ASAS domains at Week 16 were transitioned to 30 mg apremilast tablets BID and continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
- Apremilast 30 mg /Apremilast 30 mg Second Escape (SE): Participants initially randomized to 30 mg apremilast tablets BID who did not have at least 20% improvement or ≥ 1 unit improvement from baseline in 2 out of 4 of the ASAS domains from baseline at Week 24 continued to receive 30 mg apremilast tablets BID (second escape) for up to 4.5 years in the long-term extension phase.
- Apremilast 20 mg/Apremilast 30 mg SE: Participants initially randomized to 20 mg apremilast tablets BID who did not have at least 20% improvement or ≥ 1 unit improvement from baseline in 2 out of 4 of the ASAS domains at Week 24 were transitioned to 30 mg apremilast tablets BID (second escape) and continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the long-term extension phase.
Period: Placebo-controlled Phase (Week 0-24)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 30 mg Early Escape (EE) | Placebo/Apremilast 30 mg Crossover (XO) | Apremilast 30 mg /Apremilast 30 mg EE | Apremilast 20 mg /Apremilast 30 mg EE | Apremilast 30 mg /Apremilast 30 mg Second Escape (SE) | Apremilast 20 mg/Apremilast 30 mg SE
Started | 164 | 163 | 163 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 164 | 163 | 163 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 150 | 151 | 144 | 0 | 0 | 0 | 0 | 0 | 0
Early Escape at Week 16 | 51 (One participant who escaped early did not complete Week 24) | 49 | 49 (One participant who escaped early did not complete Week 24) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 145 (Completed = participants who completed the Placebo-controlled Phase) | 147 (Completed = participants who completed the Placebo-controlled Phase) | 138 (Completed = participants who completed the Placebo-controlled Phase) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 19 | 16 | 25 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 7 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase (Weeks 24 to 52)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 30 mg Early Escape (EE) | Placebo/Apremilast 30 mg Crossover (XO) | Apremilast 30 mg /Apremilast 30 mg EE | Apremilast 20 mg /Apremilast 30 mg EE | Apremilast 30 mg /Apremilast 30 mg Second Escape (SE) | Apremilast 20 mg/Apremilast 30 mg SE
Started (9 participants who completed Week 24 did not continue in the extension phase.) | 0 | 74 | 65 | 47 | 91 | 48 | 48 | 25 | 23
Completed | 0 | 69 | 61 | 41 | 85 | 43 | 43 | 22 | 21
Not Completed | 0 | 5 | 4 | 6 | 6 | 5 | 5 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 6 | 3 | 2 | 5 | 1 | 2
Not completed — Non-compliance study drug | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Period: Long-Term Extension Phase Weeks 52-260
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 30 mg Early Escape (EE) | Placebo/Apremilast 30 mg Crossover (XO) | Apremilast 30 mg /Apremilast 30 mg EE | Apremilast 20 mg /Apremilast 30 mg EE | Apremilast 30 mg /Apremilast 30 mg Second Escape (SE) | Apremilast 20 mg/Apremilast 30 mg SE
Started (24 participants who completed Week 52 did not continue in the Week 52-260 study period) | 0 | 66 | 61 | 35 | 81 | 39 | 38 | 21 | 20
Completed | 0 | 40 | 41 | 22 | 50 | 22 | 20 | 12 | 10
Not Completed | 0 | 26 | 20 | 13 | 31 | 17 | 18 | 9 | 10
Not completed — Adverse Event | 0 | 5 | 2 | 2 | 6 | 2 | 2 | 3 | 1
Not completed — Lack of Efficacy | 0 | 4 | 6 | 7 | 10 | 7 | 4 | 2 | 4
Not completed — Noncomplinace with Study Drug | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 11 | 11 | 1 | 12 | 7 | 5 | 3 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Miscellaneous | 0 | 5 | 1 | 2 | 0 | 1 | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified Intent to Treat (mITT) population included all participants who were randomized and received at least one dose of investigational product (IP); Five participants did not have a baseline SF-36 Physical Component Summary score.
Groups:
- Apremilast 30 mg: Participants initially randomized to 30 mg apremilast tablets BID in the 24-week placebo-controlled phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 164 | 163 | 163 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.89) | 45.2 (11.90) | 44.8 (11.75) | 44.7 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 56 | 138
  Male | 124 | 121 | 107 | 352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 1 | 7
  Not Hispanic or Latino | 158 | 159 | 162 | 479
  Unknown or Not Reported | 1 | 3 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Black or African American | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 158 | 154 | 158 | 470
  Other | 1 | 2 | 3 | 6
  Missing | 1 | 3 | 0 | 4
Duration of Ankylosing Spondylitis (Lower Back Pain and Stiffness) [Mean (Standard Deviation); unit: years] | 10.40 (10.375) | 11.06 (11.302) | 10.32 (9.887) | 10.60 (10.521)
Duration of Ankylosing Spondylitis [Count of Participants; unit: Participants]
  ≤ 2 years | 41 | 48 | 40 | 129
  >2 to ≤ 5 years | 29 | 23 | 26 | 78
  >5 to ≤ 10 years | 33 | 29 | 33 | 95
  >10 years | 61 | 63 | 64 | 188
Baseline Bath Ankylosing Spondylitis Functional Index (BASFI) Score (0 - 10 NRS) [Mean (Standard Deviation); unit: Units on a Scale] — The BASFI is a composite score based on a self-administered survey of 10 questions using a 0 to 10 unit numerical rating scale (NRS) that assesses the degree of mobility and functional ability. The survey consists of 8 questions regarding function in AS and the last 2 reflect the ability to manage everyday life. The patient marks a box with an X on a 0 to 10 unit NRS for 10 questions; the left-hand box of 0 = easy; the right-hand box = impossible. The resulting 0 to 100 score is divided by 10 to give a final 0 to 10 BASFI score. A higher score correlates to reduced functional ability.
  Units on a Scale | 5.76 (2.194) | 5.75 (2.061) | 5.65 (2.100) | 5.72 (2.115)
Baseline Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score (0 - 10 NRS) [Mean (Standard Deviation); unit: Units on a Scale] — The BASDAI is a composite score based on a self-administered survey of 6 questions using a 0 to 10 unit NRS that assesses for 5 major symptoms of AS: fatigue; spinal pain; peripheral joint pain/swelling; areas of localized tenderness; morning stiffness severity upon wakening; morning stiffness duration upon wakening. To give each of the 5 symptoms equal weighting, the mean of the 2 scores relating to morning stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 to 10 BASDAI score. A score of 4 or greater is considered to be indicative of active AS disease.
  Units on a Scale | 6.45 (1.319) | 6.46 (1.352) | 6.37 (1.357) | 6.42 (1.341)
Baseline Bath Ankylosing Spondylitis Metrology Index (BASMI)-Linear Score (0 - 10 NRS) [Mean (Standard Deviation); unit: Units on a Scale] — The BASMI-Linearis designed to assess axial status (ie, cervical, dorsal and lumbar spine, hips, and pelvic soft tissue) and to define clinically significant changes in spinal movement. 5 dimensions of movement (lateral lumbar flexion, tragus to wall, forward lumbar flexion, maximal intermalleolar distance, and cervical rotation) were measured and normalized on 0 to 10 unit NRS. The average of these scores is the total BASMI score, with a higher value indicating more severe limitation in spinal mobility. Population: Three participants did not have baseline BASMI data.
  Units on a Scale
    number analyzed (Participants) | 163 | 163 | 161 | 487
    (all) | 4.36 (1.608) | 4.63 (1.721) | 4.41 (1.700) | 4.47 (1.678)
Baseline Ankylosing Spondylitis Quality of Life (ASQoL) Summary Score (0-18) [Mean (Standard Deviation); unit: Units on a Scale] — The ASQoL is a validated disease specific patient reported outcomes instrument to assess the impact of ankylosing spondylitis on the QoL of individuals with emphasis on the ability of the person to fulfill his or her needs. It consisted of 18 items requesting a yes (score=1) or no (score=0) response to questions related to the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. The summary score ranges 0-18 with higher scores indicating worse quality of life. Population: Four participants did not have a baseline ASQoL score.
  Units on a Scale
    number analyzed (Participants) | 164 | 162 | 160 | 486
    (all) | 9.10 (4.639) | 8.38 (4.548) | 8.62 (4.935) | 8.50 (4.738)
Baseline Physical Component Summary Score of Medical Outcome Study Short Form 36-Item Survey [Mean (Standard Deviation); unit: Units on a Scale] — The SF- 36 is a self-administered instrument that measures the impact of disease and consists of 36 questions in 8 domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Two overall summary scores can also be obtained-a Physical Component Summary score (PCS) and a Mental Component Summary score (MCS). The PCS and MCS scores are transformed to have a mean of 50 and standard deviation of 10, with higher scores indicating better health. Scale scores range from 0 to 100, with higher scores indicating better health. Population: Five participants did not have a baseline SF-36 Physical Component Summary score.
  Units on a Scale
    number analyzed (Participants) | 164 | 162 | 159 | 485
    (all) | 32.57 (7.821) | 31.89 (8.561) | 32.16 (8.846) | 32.20 (8.402)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society 20 (ASAS 20) Response at Week 16
Description: ASAS 20 was defined as achieving an improvement from baseline of ≥ 20% and ≥ 1 unit in at least 3 of 4 ASAS domains on a scale of 0 to 10 units and no worsening from baseline of ≥ 20% and ≥ 1 unit in the remaining ASAS domain on a scale of 0 to 10 units. The 4 ASAS domains are:
  1. Patient Global Assessment of Disease (0 - 10 unit Numerical Rating Scale [NRS]); participant marks a box with an X on a 0 - 10 unit NRS; the left-hand box of 0 = not active and the right-hand box = very active
  2. Total Back Pain (0 to 10 unit NRS); participant marks a box with an X on a 0 - 10 unit NRS; the left-hand box of 0 = "no pain" and the right-hand box = "most severe pain"
  3. Function (Bath AS Functional Index [BASFI] NRS 0 - 10 unit); participant provides a self-administered survey of 10 questions assessing for degree of mobility and functional ability
  4. Inflammation domain is determined by the mean of 2 Bath AS Disease Activity Index NRS Questions #5 and #6 for morning stiffness) (0 - 10 unit)
Time Frame: Baseline and Week 16
Population: The mITT population included participants who were randomized and received at least one dose of investigation product (IP). Participants who discontinued early due to lack of efficacy were counted as nonresponders, and last observation carried forward (LOCF) imputation was used for participants who discontinued for other reasons.
Measure: Number; unit: Percentage of Participants
Groups:
- Apremilast 20 mg: Participants initially randomized to 20 mg apremilast tablets BID in the 24-week placebo-controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 163 | 163
Percentage of Participants | 36.6 | 35.0 | 32.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.4383, Cochran-Mantel-Haenszel; 2 sided p-value was based on CMH test adjusting for C-reactive protein (CRP) category and baseline BASDAI score category; Risk Difference (RD) = -4.1, 95% CI 2-sided [-14.3 to 6.2] — Adjusted difference is the weighted average of the treatment differences across the 4 strata of screening CRP category and baseline BASDAI score category with the Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.7427, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-12.0 to 8.5] — Adjusted difference in proportions is the weighted average of the treatment differences across the 4 strata of screening CRP category and baseline BASDAI score category with the Cochran-Mantel-Haenszel weights

2. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 24
Description: The BASFI is a composite score based on a self-administered survey of 10 questions using a 0 to 10 unit numerical rating scale (NRS) that assesses the degree of mobility and functional ability. The survey consists of 8 questions regarding function in AS and the last 2 reflect the ability to manage everyday life. The patient marks a box with an X on a 0 to 10 unit NRS for 10 questions; the left-hand box of 0 = easy; the right-hand box = impossible. The resulting 0 to 100 score is divided by 10 to give a final 0 to 10 BASFI score. The overall score is the mean of the 10 items and ranges from 0 to 10. A higher score correlates to reduced functional ability.
Time Frame: Baseline and Week 24
Population: The mITT population included those who were randomized and received at least one dose of IP. Missing data were imputed as baseline carried forward for participants who escaped early or discontinued early (prior to Week 24) due to lack of efficacy and LOCF for other early discontinuations
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 162 | 163 | 160
Units on a Scale | -0.94 (0.136) | -1.11 (0.137) | -0.99 (0.138)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.8032, ANCOVA; Based on an ANCOVA model for change from baseline with treatment group, CRP and baseline BASDAI score as factors and baseline value as covariate; LS Mean Difference = -0.05, 95% CI 2-sided [-0.41 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3624, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.17, 95% CI 2-sided [-0.53 to 0.19]

3. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 24
Description: The BASDAI is a composite score based on a participant self-administered survey of six questions measured using a 0 to 10 unit numerical rating scale (NRS) that assessed the participants' five major symptoms of AS: 1) fatigue; 2) spinal pain; 3) peripheral joint pain/swelling; 4) areas of localized tenderness; 5a) morning stiffness severity upon wakening; 5b) morning stiffness duration upon wakening. The participant was asked to mark the box with an X on a 0 to 10 unit NRS for each of the 6 questions. To give each of the five symptoms equal weighting, the mean of the two scores relating to morning stiffness was taken. The resulting 0 to 50 score was divided by 5 to give a final 0 to 10 BASDAI score. A BASDAI score of 4 or greater was considered to be indicative of active AS disease.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 162 | 160
Units on a Scale | -1.21 (0.136) | -1.30 (0.136) | -1.18 (0.137)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.8618, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.03, 95% CI 2-sided [-0.33 to 0.40]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.6262, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.09, 95% CI 2-sided [-0.45 to 0.27]

4. Secondary Outcome: Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society 20 (ASAS) Response at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 163 | 163
Percentage of Participants | 31.7 | 36.2 | 33.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.6958, Cochran-Mantel-Haenszel; 2 sided p-value was based on the CMH test adjusting for C-reactive protein (CRP) category and baseline BASDAI score category; Risk Difference (RD) = 2.0, 95% CI 2-sided [-8.1 to 12.2] — Adjusted difference is the weighted average of the treatment differences across the 4 strata of screening CRP category and baseline BASDAI score category with the Cochran-Mantel-Haenszel weights
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.4051, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-5.8 to 14.5] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in the Ankylosing Spondylitis Quality of Life (ASQoL) Summary Score at Week 24
Description: The ASQoL is a validated disease specific patient reported outcomes instrument to assess the impact of ankylosing spondylitis on the quality of life of individuals with emphasis on the ability of the person to fulfill his or her needs. It consisted of 18 items requesting a yes (score=1) or no (score=0) response to questions related to the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. The summary score ranges 0-18 with higher scores indicating worse quality of life.
Time Frame: Baseline and Week 24
Population: The mITT included those who were randomized and received at least one dose of IP. Missing data were imputed as baseline carried forward for participants who escaped early or discontinued early (prior to Week 24) due to lack of efficacy and LOCF for other early discontinuations.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 160 | 161 | 156
Units on a Scale | -1.77 (0.278) | -1.50 (0.278) | -1.52 (0.281)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.5126, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.25, 95% CI 2-sided [-0.49 to 0.99]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.4624, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.28, 95% CI 2-sided [-0.46 to 1.01]

6. Secondary Outcome: Change From Baseline in the Physical Component Summary Score (PCS) of Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) at Week 24
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) was a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores (based on US general population with mean of 50 and standard deviation of 10) were used in analyses. Higher scores indicate a higher level of functioning. The PCS encompasses physical functioning, role-physical, and bodily pain, as well as general health and vitality. A positive change from baseline score indicates an improvement
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 160 | 161 | 155
Units on a Scale | 3.50 (0.553) | 3.46 (0.551) | 3.79 (0.559)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.6997, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.29, 95% CI 2-sided [-1.18 to 1.76]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.9587, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-1.50 to 1.42]

7. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index-Linear (BASMI-Linear) at Week 24
Description: The BASMI-Linear was designed to assess axial status (ie, cervical, dorsal and lumbar spine, hips, and pelvic soft tissue) and to define clinically significant changes in spinal movement. Five dimensions of movement (lateral lumbar flexion, tragus to wall, forward lumbar flexion, maximal intermalleolar distance, and cervical rotation) were measured and normalized on 0 to 10 unit NRS. The average of these scores was the total BASMI score, ranging from 0-10 with higher values indicating more severe limitation in spinal mobility.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 162 | 158
Units on a Scale | -0.19 (0.042) | -0.16 (0.043) | -0.13 (0.043)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.3307, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.06, 95% CI 2-sided [-0.06 to 0.17]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.5938, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.03, 95% CI 2-sided [-0.08 to 0.14]

8. Secondary Outcome: Change From Baseline in the Radiographic Score Using the Modified Stoke Ankylosing Spondylitis Spine Score (m-SASSS) at Week 104 and Week 260
Description: The Modified Stoke Ankylosing Spondylitis Spine Score is a scoring method used to determine the amount or degree of ankylosing spondylitis disease that is in the spine based on x-ray radiographs of the spine. The m-SASSS scores 0-3.
  0 = No abnormality, 1 = Erosion, Sclerosis or Squaring, 2 = Syndesmophyte, 3 = Total bony Bridging at each Site. An increase in the m-SASSS indicated a worsening of AS disease.
Time Frame: Baseline to Week 104 and 260
Population: The radiograph subset analysis population included randomized participants who received at least one dose of IP and had at least a baseline radiograph available. Includes apremilast participants as treated who had a baseline and at least one post-baseline score. Missing scores were imputed using the LOCF.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Apremilast 20 mg: Participants initially randomized to 20 mg apremilast tablets BID in the 24-week placebo-controlled phase, and continued to receive apremilast 20 mg or 30 mg during weeks 24 to 260.
- Apremilast 30 mg: Participants initially randomized at Week 0 to 30 mg apremilast tablets BID in the 24-week placebo-controlled phase, and continued to receive apremilast 30 mg during weeks 24 to 260.
- Placebo/Apremilast 30 mg: Participants who initially received placebo tablets BID during the placebo controlled phase were transitioned to 30 mg apremilast tablets BID either at Week 16 or Week 24 through to Week 260.
- Apremilast 20 mg/ Apremilast 30 mg: Participants who were initially randomized to 20 mg apremilast tablets BID at Week 0 and transitioned to 30 mg apremilast tablets BID at either Week 16 or Week 24 through to Week 260.
- Apremilast 20 mg/Apremilast 20 mg: Participants who were initially randomized to receive 20 mg apremilast PO BID at Week 0 and continued to receive 20 mg apremilast PO BID through to Week 260 without the transition to 30 mg apremilast PO BID.
Arm/Group | Apremilast 20 mg | Apremilast 30 mg | Placebo/Apremilast 30 mg | Apremilast 20 mg/ Apremilast 30 mg | Apremilast 20 mg/Apremilast 20 mg
Number analyzed (Participants) | 83 | 84 | 79 | 35 | 48
Units on a Scale
  Week 104: number analyzed (Participants) | 81 | 81 | 74 | 35 | 46
  Week 104 | 0.99 (3.018) | 0.65 (2.453) | 0.98 (3.768) | 0.82 (2.435) | 1.12 (3.417)
  Week 260 | 3.14 (8.292) | 1.79 (6.997) | 1.92 (7.363) | 2.21 (5.959) | 3.83 (9.652)

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Placebo Controlled Phase
Description: A TEAE was an adverse event (AE) with a start date on or after the date of the first dose of IP and no later than 28 days after the last dose of IP for participants who discontinued early. A serious AE = results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect; or constitutes an important medical event. The severity of AEs was assessed based on the following scale: Mild = asymptomatic or mild symptoms, clinical or diagnostic observations only; Moderate = symptoms cause moderate discomfort; Severe = symptoms causing severe pain discomfort.
Time Frame: From Week 0 to Week 24; the median duration of exposure was 23.57 weeks for the placebo arm, 23.71 weeks for the apremilast 20 mg arm and 24.00 weeks for the apremilast 30 mg arm.
Population: Safety population includes all participants who were randomized and received at least one dose of IP. Includes data through Week 16 for placebo-treated and apremilast 20 mg BID treated participants who escaped early and data up to Week 24 for all other participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 163 | 163
Participants
  Any Treatment Emergent Adverse Event | 83 | 91 | 88
  Any Drug-related TEAE | 24 | 44 | 51
  Any Severe TEAE | 0 | 2 | 5
  Any Serious TEAE | 1 | 3 | 6
  Any Serious Drug-related TEAE | 0 | 0 | 3
  Any TEAE Leading to Drug Interruption | 14 | 13 | 14
  Any TEAE Leading to Drug Withdrawal | 7 | 11 | 13
  Any TEAE Leading to Death | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Apremilast Exposure Period
Description: as for outcome 9
Time Frame: Week 0 to week 260; overall mean duration of exposure to apremilast 20 mg and 30 mg BID was 160.96 weeks
Population: Apremilast Subjects as Treated (AAT) were those who received at least 1 dose of apremilast at any time during the study. Participants were included in the treatment group corresponding to the apremilast dosing regimen they actually received, irrespective of the treatment group to which they were randomized or re-randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast 20 mg: Participants who received 20 mg apremilast tablets BID only in the study. This also includes participants who initially received APR 20 BID and switched to APR 30 BID treatment. Only the TEAEs that occurred during the 20 mg apremilast BID dose were included.
- Apremilast 20/30 mg: Participants who initially received 20 mg apremilast tablets BID at Week 0 who escaped to 30 mg apremilast BID. Only the TEAEs that occurred during the apremilast 30 mg BID dose were included.
- Apremilast 30 mg: Participants initially randomized to 30 mg apremilast tablets BID at Week 0 and participants who received placebo at Week 0 who escaped to 30 mg apremilast BID. Only the TEAEs that occurred during the APR 30 mg BID dose were included.
Arm/Group | Apremilast 20 mg | Apremilast 20/30 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 72 | 305
Participants
  Any Treatment Emergent Adverse Event | 114 | 47 | 239
  Any Severe TEAE | 5 | 8 | 23
  Any Serious TEAE | 12 | 8 | 41
  Any TEAE Leading to Drug Interruption | 22 | 11 | 51
  Any TEAE Leading to Drug Withdrawal | 18 | 4 | 34
  Any TEAE Leading to Death | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs were reported for the placebo-controlled phase from Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants. AEs were reported for the apremilast (APR) exposure period from Week 0 to Week 260, irrespective of when the APR started (Week 0, 16 or 24). The median duration of treatment was 24, 163, and 216 weeks in the Apremilast 20 mg, Apremilast 20/30 mg and Apremilast 30 mg treatment groups respectively.
Groups:
- Placebo (Weeks 0-24) Placebo-Controlled Phase: Participants randomized to placebo tablets twice daily (BID) in the 24-week placebo-controlled phase.
- Apremilast 20 mg BID (Weeks 0-24) Placebo-Controlled Phase: Participants initially randomized to 20 mg apremilast tablets (APR) BID in the 24-week placebo-controlled phase.
- Apremilast 30 mg BID (Weeks 0-24) Placebo-Controlled Phase: Participants initially randomized to 30 mg apremilast tablets BID in the 24-week placebo-controlled phase.
- Apremilast 20 mg BID (APR Exposure Period): Participants who received 20 mg apremilast tablets BID only in the study. This also includes participants who initially received APR 20 BID and switched to APR 30 BID treatment.
  Only the TEAEs that occurred during the 20 mg apremilast BID dose were included.
- Apremilast 20/30 mg BID (APR Exposure Period): Participants who initially received 20 mg apremilast tablets BID at Week 0 who escaped to 30 mg apremilast BID. Only the TEAEs that occurred during the 20 mg apremilast BID dose were included.
- Apremilast 30 mg BID (APR Exposure Period): Participants initially randomized to 30 mg apremilast tablets BID at Week 0 and participants who received placebo at Week 0 who escaped to 30 mg apremilast tablets BID. Only the TEAEs that occurred during the 30 mg apremilast BID dose were included.
Arm/Group | Placebo (Weeks 0-24) Placebo-Controlled Phase | Apremilast 20 mg BID (Weeks 0-24) Placebo-Controlled Phase | Apremilast 30 mg BID (Weeks 0-24) Placebo-Controlled Phase | Apremilast 20 mg BID (APR Exposure Period) | Apremilast 20/30 mg BID (APR Exposure Period) | Apremilast 30 mg BID (APR Exposure Period)
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/163 | 0/163 | 0/163 | 1/72 | 1/305
Serious Adverse Events (participants affected / at risk) | 1/164 | 3/163 | 6/163 | 12/163 | 8/72 | 41/305
Other Adverse Events (participants affected / at risk) | 37/164 | 58/163 | 57/163 | 82/163 | 38/72 | 168/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-24) Placebo-Controlled Phase (N=164) | Apremilast 20 mg BID (Weeks 0-24) Placebo-Controlled Phase (N=163) | Apremilast 30 mg BID (Weeks 0-24) Placebo-Controlled Phase (N=163) | Apremilast 20 mg BID (APR Exposure Period) (N=163) | Apremilast 20/30 mg BID (APR Exposure Period) (N=72) | Apremilast 30 mg BID (APR Exposure Period) (N=305)
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Device failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infected bites (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-24) Placebo-Controlled Phase (N=164) | Apremilast 20 mg BID (Weeks 0-24) Placebo-Controlled Phase (N=163) | Apremilast 30 mg BID (Weeks 0-24) Placebo-Controlled Phase (N=163) | Apremilast 20 mg BID (APR Exposure Period) (N=163) | Apremilast 20/30 mg BID (APR Exposure Period) (N=72) | Apremilast 30 mg BID (APR Exposure Period) (N=305)
Iridocyclitis (Eye disorders) | 0 | 1 | 1 | 2 | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 9 | 7 | 1 | 16
Diarrhoea (Gastrointestinal disorders) | 7 | 22 | 17 | 26 | 4 | 38
Frequent bowel movements (Gastrointestinal disorders) | 2 | 2 | 3 | 3 | 4 | 3
Nausea (Gastrointestinal disorders) | 7 | 10 | 14 | 13 | 6 | 28
Bronchitis (Infections and infestations) | 1 | 4 | 2 | 8 | 6 | 10
Nasopharyngitis (Infections and infestations) | 6 | 9 | 7 | 25 | 10 | 55
Sinusitis (Infections and infestations) | 1 | 2 | 1 | 7 | 5 | 10
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 8 | 17 | 8 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 6 | 4 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 5 | 4 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 4 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 4 | 5
Headache (Nervous system disorders) | 8 | 9 | 16 | 11 | 5 | 28
Hypertension (Vascular disorders) | 4 | 4 | 6 | 6 | 2 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally sixty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.